CLINICAL TRIAL: NCT06911359
Title: The Effect of Non-steroidal Anti-inflammatory Drug (NSAID) Use on the Efficacy of Dextrose Prolotherapy in the Treatment of Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: The Effect and Safety of Anti-inflammatories and Dextrose Prolotherapy Injections in Treating Knee Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDG20230042H
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis (OA)
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ibuprofen group (Active Comparator)
  Interventions: Drug: Participants are given Ibuprofen 400 mg to take for 7 days on the day they receive a dextrose prolotherapy (DPT) injection. These procedures are repeated every 3-5 weeks for a total of 3 times.
- Placebo group (Placebo Comparator)
  Interventions: Drug: Participants are given a placebo to take for 7 days on the day they receive a dextrose prolotherapy (DPT) injection. These procedures are repeated every 3-5 weeks for a total of 3 times.

INTERVENTIONS:
Drug: Participants are given Ibuprofen 400 mg to take for 7 days on the day they receive a dextrose prolotherapy (DPT) injection. These procedures are repeated every 3-5 weeks for a total of 3 times. — The other group is given a placebo when they receive their dextrose prolotherapy (DPT) injection
  Arms: Ibuprofen group
Drug: Participants are given a placebo to take for 7 days on the day they receive a dextrose prolotherapy (DPT) injection. These procedures are repeated every 3-5 weeks for a total of 3 times. — The other group is given Ibuprofen when they receive their dextrose prolotherapy (DPT) injection
  Arms: Placebo group

SUMMARY:
Our purpose is to expand upon the results of the pilot study performed at David Grant Medical Center (DGMC) which showed that concomitant non-steroidal NSAID use in adults with knee osteoarthritis (OA) undergoing a three-shot dextrose prolotherapy (DPT) injection series did not negate the efficacy of DPT. Additionally, it showed that giving both treatments simultaneously is safe and efficacious. The small sample size and design of the pilot study limited the conclusions that can be drawn on the concomitant use of non-steroidal anti-inflammatory drugs (NSAIDs) during DPT treatment.

This is a double-blinded, randomized, controlled trial that includes a subject population of males and females between the ages of 45-75 years who are DoD beneficiaries empaneled at DGMC with a history of chronic, symptomatic knee osteoarthritis in one or both knees, that meet study criteria.

Participants will have study inclusion/exclusion and knee films (within the past 2 years) reviewed by a study investigator to confirm eligibility to participate in the study. Eligible participants will be consented then randomized into treatment groups (ibuprofen, placebo) by the pharmacy. Participants will provide a baseline assessment of pain and dysfunction using the Numeric Pain Rating Scale (NPRS) and Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaires. Participants will then have a series of three injections of 4mL of 25% dextrose mixed with 1% lidocaine into the knee under ultrasound guidance, performed at 0, 4 and 8 weeks (+/- 1 week) in addition to a 7-day supply of the study drug (ibuprofen, placebo) at these time points. NPRS and KOOS scores will be collected at 0, 4, 8 and 12 weeks. During the study period, participants will be counseled to avoid oral analgesics (other than what has been prescribed for them as part of the study) including NSAIDs, acetaminophen, or opioids, in addition to other procedures to treat their knee pain to include other injections, acupuncture, physical therapy, and surgery.

The primary outcome is to determine the effect of concomitant oral ibuprofen vs. placebo use on intra-articular knee injections using hypertonic dextrose and the determine the short and long-term outcomes in each treatment group (ibuprofen, placebo) using the NPRS and KOOS questionnaires to assess pain and function.

ELIGIBILITY:
Inclusion Criteria:

* Must be DoD Healthcare beneficiaries empaneled at DGMC
* Adults aged 45-75 years with a clinical diagnosis of Knee OA (either unilateral or bilateral) based on clinical and radiographic criteria as defined by the American College of Rheumatology (Altman 1987)
* Knee radiographs (within 2 years of start date) with Kellgren-Lawrence classification of 2-3
* Moderate to severe Knee pain for at least 3 months defined as a score of ≥4 using the NPRS (0-10) in response to the question "What is the average level of your left/ right knee pain in the past 3 months?"
* English speaking
* Not pregnant
* Not breastfeeding
* No allergy to dextrose, lidocaine, or sulfite

Exclusion Criteria:

* Previous knee replacement surgery
* Previous meniscus repair/debridement surgery or chondral replacement surgery
* Any intra-articular injection including steroid, prolotherapy or platelet rich plasms within the previous 3 months
* Significant effusion as defined by a ballotable patella
* Pregnancy or breastfeeding
* Current/ongoing medical problems obtained from chart review contraindicating NSAID use to include chronic kidney disease stage II or higher, acute interstitial nephritis, coronary artery disease requiring percutaneous coronary intervention (PCI) or bypass surgery; Major Adverse Coronary Event (MACE), body mass index (BMI) ≥40, inflammatory arthropathy (gouty arthritis, psoriatic arthritis, or septic arthritis), history of GI bleed.
* Non-English speaking
* Allergy to dextrose, lidocaine, or sulfite

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Injury in Osteoarthritis (KOOS) questionnaire scores | From enrollment to the end of treatment at 12 weeks
  The KOOS questionnaire consist of a total of 23 items divided (unequally) among 5 subscales. The subscales include pain (5 items), symptoms (4 items), activities of daily living (ADL) (9 items), sport/recreation (3 items), and quality of life (QoL) (2 items). Each item is scored on a scale of 0-4. Zero is assigned to "never", "none," and "not at all" responses. Four is assigned to "always", "extreme," "totally," and "constantly" responses. Calculate mean scores for each subscale by adding the scores for each item (in the subscale) then dividing it by the total number of items (in the subscale). Then multiply the calculated mean scores (for each subscale) by 100, divide it by 4, then subtract it from 100. Total subscale scores range from 0 -100. 0 indicates extreme problems and 100 indicates no problems.
Change in Numeric Pain Rating Scale (NPRS) scores | From enrollment to the end of treatment at 12 weeks
  The NPRS is a 1-item questionnaire assessing pain severity using a number which describes the level of knee pain over the last 24 hours. Participants are to put an "X" on a linear scale from 0-10. Zero (0) is no pain and 10 is the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Kim, MD, Principal Investigator — David Grant USAF Medical Center
Locations (1):
- David Grant USAF Medical Center, Travis AFB, California, United States